CLINICAL TRIAL: NCT03843814
Title: A Pilot Study Using Amide Proton Transfer (APT) Magnetic Resonance Imaging to Distinguish Tumor Bearing Cancerous Tissue From Normal Tissue in Patients With Glioma.
Brief Title: Pilot Study Using Amide Proton Transfer Magnetic Resonance Imaging Distinguishing Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Imaging results were not sufficient or of good quality; therefore, we will not move further with the project.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1439; IRB00032866 (Other: JHMIRB)
Record Dates: First submitted 2014-09-18; First posted 2019-02-18 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Gliosarcoma; Glioma
Keywords: MRI (Magnetic Resonance Imaging) of the brain; Amide Proton Transfer (APT); Diffuse Weighted Imaging (DWI)
MeSH Terms: conditions — Gliosarcoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- APT MRI (Experimental): Participants will have the standard MRI of the brain that is performed for radiation planning for brain tumors.
  1. Addition of the additional MRI sequences to the standard MRI before radiation therapy. This typically adds 10-15 minutes to the length of the scan.
  2. An additional MRI scan to be scheduled during one of the final five radiation treatment days that would not otherwise occur. There will be no contrast injection as part of this second scan. This may typically take 40-45 minutes.
  3. Collection of information about participants' tumor, including copies of their MRIs and later outcome of treatment.
  Interventions: Procedure: APT MRI

INTERVENTIONS:
Procedure: APT MRI

SUMMARY:
This research is being done to study the pattern of changes in various parts of the magnetic resonance imaging (MRI) studies that patients have done to help plan their radiation therapy and to evaluate the effects of therapy.

The MRI of the brain is one of the major ways a participant's doctors determine how to treat a participant's tumor and if the participant's tumor is growing or not. In this study the investigators want to learn if new sequences added to the MRI that the investigators are already getting to guide partipants' radiation treatment can be analyzed to help make better treatment decisions. MRI sequences that examine the composition and structure of the tissues in the brain in a different way will be obtained. These are called called Amide Proton Transfer (APT) and Diffusion Weighted MRI.

These scans will first be performed at the time of participants' radiation plannings scan done before treatment and near the end of the course of radiation treatments. This will allow the study team to investigate if there are changes in these sequences before radiation treatment and to see if using these MRI studies will allow us to better plan radiation treatments for patients in the future. This pre-treatment scan will be done at the same time as participants' standard radiation planning MRI, but will cause the scan to take longer. Participants will also have an extra MRI during one of the last 5 days of the planned 28-33 radiation treatments that are standardly used. This additional scan will not include administration of injected contrast agents, and would occur on a day when participants are also coming in for radiation. This scan will be compared with the first scan. The investigators will determine whether these changes may predict later long term outcome of treatment for patients. Patients who enroll in this study will get all of the standard therapy they would get for their tumor whether or not they participate in this study. There is no extra or different therapy given.

The investigators anticipate that the radiation treatment volumes created using APT will largely overlap with the conventional plan but will be distinct at the margins. Disease failure is more likely to occur in areas with APT abnormalities suggestive of active tumor. In patients that have failure outside the contrast enhancing area, the region of failure will be predicted by regions of increased APT activity. Current MRI sequences do not allow for prediction of regions of recurrence or progression, or distinguish between tumor, pressure, or surgical injury as the cause of FLAIR/T2 abnormalities. Disease failure is more likely to occur in areas with APT abnormalities suggestive of active tumor. In patients that have failure outside the contrast enhancing area, the region of failure will be predicted by regions of increased APT activity. Current MRI sequences do not allow for prediction of regions of recurrence or progression, or distinguish between tumor, pressure, or surgical injury as the cause of FLAIR/T2 abnormalities. Volume containing elevated APT signal may be associated with outcome (survival). In an exploratory analysis, the investigators will evaluate whether there are characteristic patterns that should be prospectively studied in a larger trial.

DETAILED DESCRIPTION:
Currently, all brain tumors are routinely evaluated using gadolinium contrast-enhanced (Gd-CE) MRI, in combination with T2-weighted or fluid-attenuated inversion recovery (FLAIR) MRI, which are used to determine the extent of tumor involvement to guide treatments, and to assess therapeutic response. However, Gd-CE only depicts disruption of the blood brain barrier and is not specific for tumor activity. Therefore, standard MRI may not be optimal in defining the true extent of tumor, defining as abnormal areas that may contain only edema related to mass effect or surgery and miss tumor extensions that do not sufficiently disrupt the blood-brain-barrier. In addition, in the setting of radiation therapy which also disrupts the blood brain barrier, it does not serve as an early marker of tumor response.

The primary goal of the current observational study is to explore whether Amide Proton Transfer (APT) imaging can better determine the extent of tumor involvement. APT signal is created by mobile cytoplasmic proteins, which are increased in malignant brain tumors and have been found in preclinical and clinical studies to be associated with a high APT weighted signal in glioma. Such imaging may provide information that may improve the ability of MR imaging to guide targeting of radiotherapy. In particular, it may (1) detect tumor bearing brain that is not contrast enhancing on the standard brain MRI scan for patients with high grade glioma and/or (2) fail to confirm tumor in areas of brain identified as abnormal on standard MRI. The investigators will also explore patterns of disease failure in patients with malignant gliomas to validate the observations, and whether such imaging may predict outcome.

Similar questions may be important in the therapy of low grade glioma, and an exploratory informational cohort of patients with this less common diagnosis will be accrued during the study period to inform decisions about whether further study is desirable.

A second APT image will be obtained during the final week of treatment for enrolled patients to determine whether changes in APT signal occur, and whether there is evidence that this may be prognostic for treatment success or failure when correlated with progression free survival and survival outcome. Currently, there is no imaging method to assess tumor response and predict outcome within the first several months as a result of the confounding effect of radiation on both the tumor and surrounding brain. In addition, standard brief apparent diffusion coefficient (ADC) MRI sequences will be performed as part of the pretreatment imaging and the end of treatment scan as an additional potential early imaging biomarker that may be a part of multiparametric assessment of response to radiotherapy as identified in preclinical studies performed at Johns Hopkins.

These first steps may form the basis for possible future studies to assess new approaches to radiation planning for patients with brain cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically Confirmed Glioma after completion of planned biopsy or resection.

   High grade glioma histologies:
   * Glioblastoma
   * High Grade or Malignant Glioma
   * Anaplastic Astrocytoma
   * Anaplastic Oligodendroglioma
   * Gliosarcoma
   * Mixture of any of the above histologies Low Grade Histologies
   * Astrocytoma
   * Grade II or low grade glioma
   * Oligodendroglioma
   * Mixtures of the above histologies
2. Plan to undergo external radiation treatment as part of therapy
3. No prior therapeutic cranial radiotherapy
4. Can safely perform clinically indicated MRI (no contraindications to MRI with Gadolinium) as determined by the standard Johns Hopkins Radiation Oncology screening procedures,

Exclusion Criteria:

1. Patients who cannot undergo MRIs.
2. Patients who are allergic to gadolinium based contrast agent
3. Patients who have cardiac pacemaker or other electronic or metal implant
4. Patients who have chronic kidney disease judged sufficient to exclude them from the clinically indicated contrast enhanced MRI.
5. Female patients who is pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Standard planning versus Amide Proton Transfer (APT) imaging planning | day 23-28 post radiation treatment
  Difference in radiation target volumes between standard MRI and Amide Proton Transfer (APT) imaging.

SECONDARY OUTCOMES:
tumor recurrence | up to 3 years
  Number of days from Day 23-28 (end of radiation) to tumor recurrence
Survival | up to 3 years
  Number of months from end of radiation therapy until death
Time to absolute change in voxels of APT and DWI (diffusion weighted imaging) signals from baseline to end of radiation treatment | Change from Baseline to Days 23-28 post-radiation treatment
  Number of days to absolute change in voxels at the end of radiation treatment.
Change in voxels of APT and DWI signals | up to 3 years or until death, whichever occurs first.
  Change in voxels of APT and DWI signal or pattern during the course of radiation treatment assessed at 3 years or until death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kleinberg, M.D., Principal Investigator — The SKCCC at Johns Hopkins
Locations (1):
- The SKCCC at Johns Hopkins, Baltimore, Maryland, United States